CLINICAL TRIAL: NCT05011903
Title: Cross-Tailoring Integrative Alcohol and Risky Sex Feedback for College Students: A Hybrid Type 1 Effectiveness-Implementation Trial
Brief Title: Integrative Alcohol and Risky Sex Feedback for College Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anne E Ray (Other)
Collaborators: University of North Texas Health Science Center (Other); Klein Buendel, Inc. (Industry); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Anne E Ray, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 62769; R01AA028246 (NIH)
Record Dates: First submitted 2021-08-10; First posted 2021-08-18 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-10

CONDITIONS: Alcohol Drinking in College; Sexual Behavior
MeSH Terms: conditions — Alcohol Drinking in College; Sexual Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PFI+CDF with diary surveys (Experimental): Participants in this condition receive a Personalized Feedback Intervention (PFI) and Cross-tailored Dynamic Feedback (CDF) related to alcohol use and related sexual behavior. They also complete weekend diary surveys in which they are asked to self-report on weekend behaviors.
  Interventions: Behavioral: Cross-tailored Dynamic Feedback; Behavioral: Personalized Feedback Intervention
- PFI+GHI with diary surveys (Experimental): Participants in this condition receive a Personalized Feedback Intervention (PFI) related to alcohol use and related sexual behavior, and generic health information (GHI). They also complete weekend diary surveys in which they are asked to self-report on weekend behaviors.
  Interventions: Behavioral: Personalized Feedback Intervention; Behavioral: Dynamic Feedback on General Health Behaviors
- PFI-only with no diary surveys (Experimental): Participants in this condition receive a Personalized Feedback Intervention (PFI) related to alcohol use and related sexual behavior. They do not complete weekend diary surveys.
  Interventions: Behavioral: Personalized Feedback Intervention
- Control (No Intervention): Participants in this condition get no intervention and do not complete weekend diary surveys.

INTERVENTIONS:
Behavioral: Cross-tailored Dynamic Feedback — Dynamic, technology-delivered weekly feedback on weekend diary self-reports of first-year college student behavior related to alcohol use and related sexual behaviors.
  Arms: PFI+CDF with diary surveys
Behavioral: Personalized Feedback Intervention — Technology-delivered personalized feedback on first-year college student behavior related to alcohol use and related sexual behaviors.
  Arms: PFI+CDF with diary surveys; PFI+GHI with diary surveys; PFI-only with no diary surveys
Behavioral: Dynamic Feedback on General Health Behaviors — Dynamic, technology-delivered weekly feedback on weekend diary self-reports of first-year college student behavior related to general health behaviors.
  Arms: PFI+GHI with diary surveys

SUMMARY:
Alcohol misuse and related risky sexual behaviors are significant health concerns for college students. Two-thirds of students are current drinkers, at least 1 in 3 report past month heavy episodic drinking (5+ drinks in a row), and 1 in 10 report high intensity drinking (10+ drinks in a row). Increased student alcohol use and heavy drinking are linked to increased sexual activity and related risky behaviors (e.g., unprotected sex, sex with casual partners). This puts students at risk for negative health outcomes (e.g., STIs - sexually transmitted infections) and is also a pathway to sexual victimization and escalated drinking. The first few weeks of college, known as the 'red zone,' provide an opportunity to intervene at time when these behaviors increase. However, most prevention programs for college students tend to focus on student alcohol use and have little to no integration of content on the relationship between alcohol use and risky sexual behaviors. This is an important gap in the literature and a priority area for NIAAA. The research team established the short-term efficacy of a personalized feedback intervention (PFI), a gold standard intervention approach, with integrated content on alcohol and risky sexual behaviors. In this study, we propose to extend our integrated PFI to include a cross-tailored dynamic feedback (CDF) component. The CDF component will use technology to incorporate daily assessments of student behavior and provide students with dynamic weekly feedback over 12 weeks. The goal is to increase the effectiveness of the integrated PFI and to create a program that is easily implemented on college campuses.

DETAILED DESCRIPTION:
The project utilizes a multisite, hybrid type 1 effectiveness-implementation study design to (1) evaluate the impact of CDF for first-year college students and (2) identify implementation factors critical to its success to facilitate future scale-up in campus settings. The first aim is to conduct a multi-level stakeholder-engaged adaptation of the integrated alcohol and risky sex PFI through the development and inclusion of CDF. The second aim is to conduct a randomized controlled trial (RCT) of the enhanced intervention (PFI+CDF) in a sample of 600 first-year college students. The primary hypothesis is that participants who receive the PFI+CDF intervention will report less alcohol use, fewer risky sexual behaviors, and fewer consequences relative to those who receive a PFI supplemented with generic health information at follow-up (1, 2, 3, 6, and 13 months). Participants (N=600 total, 300 per site) will be randomized to 1 of 4 groups: (1) PFI+CDF with weekend diary surveys, (2) PFI+GHI with weekend diary surveys, (3) PFI-only, no weekend diary surveys, and (4) assessment-only control, no weekend diary surveys. All participants will complete a baseline survey during the first week of the semester, be randomly assigned to condition, and complete follow-up surveys at 1, 2, 3, 6, and 13 months. This staggered design allows for comparison of the enhanced PFI+CDF relative to the PFI+GHI condition, which may be consistent with a "treatment-as-usual" comparison group (e.g., of the universities that have adopted an evidence-guided alcohol intervention program for their campus, many currently deliver commercialized alcohol-focused PFIs to incoming first-year students). Providing weekly GHI in the comparison condition allows for an equal number of "exposures" between the more intensive conditions (PFI+CDF vs. PFI+GHI), analogous to an attention control group, offering a clearer understanding of the overall impact of the PFI+CDF adaptation. The inclusion of two PFI conditions, one with weekend diary assessments and one without allows us to control for potential assessment reactivity that might result from the diary-style assessment approach. Overall, this design is intended to allow a separation of the "true" intervention effect of the CDF above and beyond the effect of assessment reactivity. The PFI-only vs. assessment-only control group comparison will provide a test of basic efficacy of the integrated PFI that has been adapted based on stakeholder feedback. The third aim seeks to identify factors critical to PFI+CDF implementation in campus settings through conducting focus groups with a subset of students from the RCT and with local and national systems-level stakeholders. The intervention has strong potential for widespread dissemination and targets a group at high risk for alcohol misuse and RSB.

ELIGIBILITY:
Inclusion Criteria:

* status as first-year college student at University of Kentucky or UNT-Denton
* 18-20 years old

Exclusion Criteria:

* the inability or unwillingness to give informed, voluntary consent to participate
* not meeting inclusion criteria
* currently in treatment to reduce alcohol or other substance use
* pregnant or planning to become pregnant

Ages: 18 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported alcohol-related sexual behavior frequency | Baseline, 1-month, 2-month, 3-months, 6-months, and 13-months
  Number of times alcohol was consumed during or before sex in the last month
Change in self-reported alcohol-related sexual behavior quantity | Baseline, 1-month, 2-month, 3-months, 6-months, and 13-months
  Number of alcoholic beverages consumed before sex in the last month
Change in self-reported alcohol-related hook-ups | Baseline, 1-month, 2-month, 3-months, 6-months, and 13-months
  Number of alcohol-related hook-ups experienced in the last month
Change in self-reported alcohol-related sexual behavior consequences | Baseline, 1-month, 2-month, 3-months, 6-months, and 13-months
  Number of alcohol-related sexual consequences experienced in the last month

SECONDARY OUTCOMES:
Change in self-reported alcohol use quantity | Baseline, 1-month, 2-month, 3-months, 6-months, and 13-months
  Typical number of drinks consumed on each day of week in the last month
Change in self-reported heavy episodic drinking | Baseline, 1-month, 2-month, 3-months, 6-months, and 13-months
  Number of heavy drinking episodes (4+ drinks female, 5+ drinks male) in the last month
Change in self-reported quantity of sex partners | Baseline, 1-month, 2-month, 3-months, 6-months, and 13-months
  Number of casual sex partners in the last month
Change in self-reported condom use | Baseline, 1-month, 2-month, 3-months, 6-months, and 13-months
  Number of times condom was used during sex in the last month

CONTACTS AND LOCATIONS:
Overall Officials: Anne E Ray, PhD, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - University of Kentucky, Lexington, Kentucky
  - University of North Texas Health Science Center at Fort Worth, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data will be available to qualified researchers after the main findings are published in a peer-reviewed journal upon request. All data sharing will comply with local, state, and federal laws and regulations, including HIPAA Privacy and Security Rules. Data will be de-identified before presentations and publications, as well as any datasets shared with qualified researchers.
Supporting Information: Study Protocol
Time Frame: To be determined.
Access Criteria: To be determined.

REFERENCES:
- [Derived] Ray AE, Mun EY, Lewis MA, Litt DM, Stapleton JL, Tan L, Buller DB, Zhou Z, Bush HM, Himelhoch S. Cross-Tailoring Integrative Alcohol and Risky Sexual Behavior Feedback for College Students: Protocol for a Hybrid Type 1 Effectiveness-Implementation Trial. JMIR Res Protoc. 2023 Mar 20;12:e43986. doi: 10.2196/43986. PMID 36716301